CLINICAL TRIAL: NCT00162617
Title: The Effect of Liberal vs. Restrictive Transfusion Strategies on Rehabilitation After Hip Fracture Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: IMK Fonden (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HHSG-RCT-03
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2006-09

CONDITIONS: Hip Fracture
Keywords: Hip fracture; Rehabilitation; Transfusion; Outcome
MeSH Terms: conditions — Hip Fractures | interventions — Erythrocyte Transfusion

INTERVENTIONS:
Drug: Red blood cell transfusion

SUMMARY:
To examine the effect of two different transfusion regimens on rehabilitation after hip fracture surgery.

DETAILED DESCRIPTION:
The effect of liberal vs restrictive transfusion regimens after hip fracture surgery is unresolved. Liberal transfusion regimens (transfusion trigger hgb. 6.25 mmol/l) leads to an increased use of blood products but may impact positively on rehabilitation outcome, a restrictive transfusion trigger (hbg. 5.0 mmol/l) saves blood products but may also impair postoperative rehabilitation and outcome. the study randomizes 120 elderly patients with hip fractures to either a restrictive or a liberal perioperative transfusion therapy and measures postoperative rehabilitation outcomes within a well defined multimodal rehabilitation regimen.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip fracture
* capable of informed consent
* independently dwelling
* able to ambulate independent of human assistance
* no active heart condition defined as no AMI within 3 months, no unstable angina or present incompensation/pulmonary oedema
* no regular transfusion demand or terminal disease.

Exclusion Criteria:

* Multiple fractures
* postop. immobilization due to to surgical reasons
* patient refusal to participate in relevant rehabilitation
* reoperation within 4. postoperative day.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120
Dates: Start 2004-01; Study Completion 2006-03

PRIMARY OUTCOMES:
Postoperative Functional mobility
Restricting factors for functional mobility

SECONDARY OUTCOMES:
Length of stay
Complications
Dizziness
Exhaustion
Haematoma (leg swelling)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, MD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Foss NB, Kristensen MT, Jensen PS, Palm H, Krasheninnikoff M, Kehlet H. The effects of liberal versus restrictive transfusion thresholds on ambulation after hip fracture surgery. Transfusion. 2009 Feb;49(2):227-34. doi: 10.1111/j.1537-2995.2008.01967.x. PMID 19389209